CLINICAL TRIAL: NCT05444569
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Study to Evaluate the Safety and Tolerability of LY3537021 When Combined With GLP-1 Receptor Agonist in Healthy Participants
Brief Title: A Study of LY3537021 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18449; J2R-MC-YAAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Healthy
MeSH Terms: interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: The study has two parts. Part A is parallel model and part B is crossover.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LY3537021 + Liraglutide (Part A) (Experimental): Liraglutide administered subcutaneously (SC) followed by liraglutide in combination with LY3537021 given SC.
  Interventions: Drug: LY3537021; Drug: Liraglutide
- Liraglutide + Placebo (Part A) (Experimental): Liraglutide administered SC followed by liraglutide in combination with placebo given SC.
  Interventions: Drug: Liraglutide; Drug: Placebo
- LY3537021 + Liraglutide & Placebo + Liraglutide (Part B) (Experimental): LY3537021 administered SC followed by liraglutide administered SC in treatment period 1.
  Placebo administered SC followed by liraglutide administered SC in treatment period 2.
  Interventions: Drug: LY3537021; Drug: Liraglutide; Drug: Placebo
- Placebo + Liraglutide & LY3537021 + Liraglutide Part B) (Experimental): Placebo administered SC followed by liraglutide administered SC in treatment period 1.
  LY3537021 administered SC followed by liraglutide administered SC in treatment period 2.
  Interventions: Drug: LY3537021; Drug: Liraglutide; Drug: Placebo

INTERVENTIONS:
Drug: LY3537021 — Administered SC.
  Arms: LY3537021 + Liraglutide & Placebo + Liraglutide (Part B); LY3537021 + Liraglutide (Part A); Placebo + Liraglutide & LY3537021 + Liraglutide Part B)
Drug: Liraglutide — Administered SC.
Drug: Placebo — Administered SC.
  Arms: LY3537021 + Liraglutide & Placebo + Liraglutide (Part B); Liraglutide + Placebo (Part A); Placebo + Liraglutide & LY3537021 + Liraglutide Part B)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3537021 when administered in combination with glucagon-like peptide (GLP-1) receptor agonist called liraglutide in treatment-naïve healthy participants. The study will include 2 parts. The study will last up to 16 and 22 weeks for part A and B, respectively which includes a screening period of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined through medical evaluation
* Participants with body weight at least 55 kilograms (kg) and body mass index (BMI) of 23.0 to 40.0 kilograms per meter squared (kg/m²)
* Males, or females who are not of childbearing potential.
* Capable of giving signed informed consent form
* Have blood pressure of less than 150/90 millimeters of mercury (mm Hg) and pulse rate of less than 100 beats per minute (bpm) (supine)

Exclusion Criteria:

* Have a significant history of current disorders capable of significantly altering the absorption, metabolism or elimination of drugs
* History of malignancy within 5 years prior to screening
* Have evidence of significant active psychiatric disorder(s)
* Have undergone any form of bariatric surgery
* Have an abnormality in the 12-lead electrocardiogram (ECG)
* Are females who are lactating

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Week 22
  A summary of TEAEs and SAEs, regardless of causality, will be reported in the Reported Adverse Events module

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No